CLINICAL TRIAL: NCT02286973
Title: Combined Administration of Intravenous and Topical Tranexamic Acid in Total Knee Arthroplasty: Is it the Most Effective Regime? A Randomized Controlled Trial.
Brief Title: Combined Administration of Intravenous and Topical Tranexamic Acid in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyun Kim, Director, Clinical Research, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1407/257-005
Record Dates: First submitted 2014-10-27; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Degenerative Arthritis
Keywords: Tranexamic acid
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Only Intravenous Group (Active Comparator): Only Intravenous Injection During Operation, 10mg/kr
  Interventions: Drug: Tranexamic Acid
- Intravenous + Topical 1g Group (Active Comparator): Intravenous Injection During Operation, 10mg/kr
  After Capsule Closure, Tranexamic acid Topical Injection 1g
  Interventions: Drug: Tranexamic Acid
- Intravenous + Topical 2g Group (Active Comparator): Intravenous Injection During Operation, 10mg/kr
  After Capsule Closure, Tranexamic acid Topical Injection 2g
  Interventions: Drug: Tranexamic Acid
- No Intravenous, Only Topical 2g Group (Active Comparator): Only Topical Injection 2g
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid

SUMMARY:
This prospective randomized controlled trial was conducted To compare the efficacy of TNA in terms of total blood loss and the allogenic transfusion rate among the three study groups; intravenous alone, combined intravenous and low dose topical TNA and combined intravenous and high dose topical TNA.

To evaluate the safety of each regimen in view of deep vein thrombosis and venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of primary osteoarthritis

Exclusion Criteria:

* patients with diagnoses other than primary OA
* patients on anticoagulation therapy
* patient with chronic renal failure
* patient with CVA Hx
* Patient with seizure Hx
* Patient with severe CHF
* Patient with acquired or congenital coagulopathy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin | baseline and 5 days
  Blood loss reduce